CLINICAL TRIAL: NCT03087032
Title: Efficacy and Safety of Liraglutide-bolus (Liraglutide Plus Prandial Insulin) Versus Glargine-bolus Therapy in Overweight / Obese Patients With Uncontrolled Type 2 Diabetes (LiraGooD)--A Multicenter Randomized Controlled Study
Brief Title: Liraglutide-bolus vs Glargine-bolus Therapy in Overweight/Obese Type 2 Diabetes Patients (LiraGooD)
Acronym: LiraGooD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYH2017-002
Record Dates: First submitted 2017-03-08; First posted 2017-03-22 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Patients; Overweight and Obesity; Hyperglycaemia (Diabetic)
Keywords: Liraglutide; Insulin Glargine; Prandial Insulin
MeSH Terms: conditions — Overweight; Obesity; Hyperglycemia | interventions — Liraglutide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide-bolus (Experimental): 'Liraglutide-bolus'(Liraglutide once-daily plus thrice-daily prandial insulin lispro). Patients will receive adding Liraglutide to prandial insulin Lispro. The starting liraglutide dose was 0.6mg/day, then 1.2mg/day after 1 week and 1.8mg/day after a further week. The dose was maintained until study completion. Dose of insulin Lispro will be instructed on a titration schedule, adjusted every 3 days.
  Interventions: Drug: Liraglutide
- Basal-bolus (Active Comparator): 'Basal-bolus' (insulin glargine once-daily plus thrice-daily prandial insulin lispro). Patients will receive adding insulin Glargine to prandial insulin Lispro.Dose of insulin will be instructed on a titration schedule, adjusted every 3 days. Patients subcutaneously self-injected once-daily at approximately the same time each day.
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: Liraglutide — Patients will receive adding Liraglutide to prandial insulin Lispro. The starting liraglutide dose was 0.6mg/day, then 1.2mg/day after 1 week and 1.8mg/day after a further week. The dose was maintained until study completion. Dose of insulin Lispro will be instructed on a titration schedule, adjusted every 3 days.
  Other Names: Victozaa; Liraglutid; Liroglutide; Liraglutidum; Liraglutide Acetate
  Arms: Liraglutide-bolus
Drug: insulin glargine — Individuals randomized to adding insulin Glargine to prandial insulin Lispro will be instructed on a titration schedule, adjusted every 3 days. Patients subcutaneously self-injected once-daily at approximately the same time each day.
  Other Names: Lantus
  Arms: Basal-bolus

SUMMARY:
The present 24-week, prospective, open-label, randomized, multicenter, parallel group trial is carried to investigate and evaluate the efficacy and safety of Liraglutide in combination with prandial insulin therapy vs insulin glargine in combination with prandial insulin therapy in overweight / obese patients with uncontrolled type 2 diabetes.

DETAILED DESCRIPTION:
An increasing number of patients with type 2 diabetes are treated with insulin. Patients with diabetes receiving intensive insulin therapy with various combinations of basal and prandial insulin can be caught in a vicious but common cycle, whereby insulin requirements increase over time, and this in turn contributes to weight gain and hypoglycemia and further increases in insulin dosing. At this stage, clinicians observe a practical limit to the efficacy of insulin titration alone on glucose-lowering and often add or continue metformin to reduce insulin resistance. Injectable glucagon-like peptide-1 receptor agonists (GLP-1 RAs), such as liraglutide, are a relatively new addition to our treatment armamentarium. These drugs improve glucose control and insulin sensitivity and contribute to weight loss. Treatment with basal insulin plus GLP-1RAs is well-established in diabetes guidelines and may be as effective as adding prandial insulin therapy. When GLP-1 RAs are started, a preemptive reduction in insulin dosage by 25% to 30% in patients with HbA1c < 9% may reduce the risk for hypoglycemia. In overweight/obese patients with uncontrolled type 2 diabetes treated with more than three oral antidiabetic drugs (OADs) or high doses of premix insulin, Is basal-prandial insulin therapy the option treatment algorithm? Such an intensification strategy carries risk of increased hypoglycaemia and weight gain, both of which are associated with worse long-term outcomes. There have no randomized, controlled trials to evaluate the efficacy and safety of GLP-1 RAs vs insulin glargine added to prandial insulin in overweight/obese patients with uncontrolled type 2 diabetes. So, the current 24-week, prospective, open-label, randomized, multicenter, parallel group trial will be preformed to assess whether Liraglutide plus prandial insulin therapy was superior to glargine plus prandial insulin therapy in overweight/obese patients with uncontrolled type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years old.
* BMI must be greater than 24 and less than 45 kg/m2
* Patients with type 2 diabetes who met the World Health Organization (who) diagnostic criteria (1999).
* Newly diagnosed type 2 diabetic patients with HbA1c ≥ 9.0%；or patients with uncontrolled type 2 diabetes (HbA1c ≥ 7.5% ) who have received at least two types of oral hypoglycemic drugs (the dose of each drug needs to reach the second largest dose or more), or only insulin (excluding basal-bolus insulin therapy), or insulin with oral hypoglycemic drugs.
* Signed informed consent.

Exclusion Criteria:

* History of pancreatic disease,
* History of medullary thyroid carcinoma
* Lipase level > 3 times above normal,
* Creatinine clearance ≤ 30 mL/min/1.73m2,
* Evidence in the last 6 months of significant heart disease or stroke, including myocardial infarction, unstable angina, coronary bypass and/or percutaneous transluminal coronary angioplasty, congestive heart failure (New York Heart Association Functional Classification III-IV), or severe ischemic heart disease.
* Preparation for pregnancy or having been in pregnancy
* Researchers believe that there are any factors that affect assessing subjects' participation in trial.
* Patients unable to cooperate in clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with HbA1c < 7.0% without experiencing hypoglycemia and without weight gain,with a superiority margin of 3% | 24 weeks
  the net difference in the proportion of patients with HbA1c < 7.0% without experiencing hypoglycemia and without weight gain is more than 3%

SECONDARY OUTCOMES:
the proportion of patients with hypoglycemia | 24 weeks
  the proportion of patients with hypoglycemia
changes in HbA1c | 24 weeks
  changes in HbA1c
changes from baseline in FPG(mmol/L) | 24 weeks
  changes from baseline in FPG(mmol/L)
changes in body weight ( kilograms) | 24 weeks
  changes in body weight( kilograms)
changes in prandial insulin dosage （per kilogram） | 24 weeks
  changes in prandial insulin dosage （per kilogram）
changes in visceral as assessed by dual x-ray absorptiometry (DXA) | 24 weeks
  changes in visceral as assessed by dual x-ray absorptiometry (DXA)
number of participants with abnormal laboratory values and/or adverse events that are related to treatment | 24 weeks
  number of participants with abnormal laboratory values and/or adverse events
changes in serum c-peptide level | 24 weeks
  changes in serum c-peptide level
changes in systolic pressure | 24 weeks
  changes in systolic pressure
changes in diastolic pressure | 24 weeks
  changes in diastolic pressure
changes in serum lipid profile | 24 weeks
  changes in serum lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Xuejun Li, MD, Principal Investigator — The first afilliated hospital of Xiamen university
Locations (1):
- The first afilliated hospital of Xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided